CLINICAL TRIAL: NCT04345055
Title: Immediate Impact of Lumbar Fascia Stretching on Hamstring Flexibility: a Randomized Clinical Trial
Brief Title: Immediate Impact of Lumbar Fascia Stretching on Hamstring Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, David Perez Cruzado, Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CONSORT
Record Dates: First submitted 2020-04-06; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Hamstring Injury
Keywords: hamstring muscles; lumbar fascia; flexibility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial treatment (Experimental): Treatment the lumbar fasciae
  Interventions: Other: Treatment of the lumbar fasciae
- Placebo group (Placebo Comparator): Introduce in a machine off
  Interventions: Other: Placebo intervention

INTERVENTIONS:
Other: Treatment of the lumbar fasciae — Treat the lumbar facial with a manual technique
  Arms: Fascial treatment
Other: Placebo intervention — Introduce in a machine off
  Arms: Placebo group

SUMMARY:
Introduction: the hamstring muscles has a great tendency to decrease its extensibility, originating a pathology with a own clinical entity, the Short Hamstring Syndrome (SHS), in addition to other problems on adjacent structures. All this present a great socioeconomic impact in the investigator's society. Various techniques have been demostrated to prduce an increase in flexibility, among which are the fascial techniques.

Objective: to evaluate the immediate efficacy of the treatment of the lumbar fascia in the flexibility of the hamstring musculature.

Methods: 41 women between 18 and 39 years old, in two groups. The experimental group received a technique of fascial stretching in the lumbar area while the control group participated in an off magnetotherapy machine. The hamstring flexibility in both lower limbs was measured by the Straight Leg Raising Test (SLR) and the Passive Popliteal Angle Test (PKE).

DETAILED DESCRIPTION:
The hamstring muscles has a great tendency to decrease its extensibility, originating a pathology with a own clinical entity, the Short Hamstring Syndrome (SHS), in addition to other problems on adjacent structures. This study aims to help improve treatment for the problem mentioned before, which can be included within a therapeutic framework to combat SHS. In recent years, investigations have been carried out that include different techniques for stretching the hamstring muscles, as well as the treatment of other structures belonging to the posterior superficial chain. Within this last section, myofascial stretching techniques have been shown to be effective both in the short and medium term. Different techniques for stretching the hamstring muscles have been carried out with the aim of increasing the flexibility of the lower back in general.

he objective is to evaluate the immediate efficacy of the treatment of the lumbar fascia in the flexibility of the hamstring musculature.

The participants are 41 women between 18 and 39 years old, in two groups. The experimental group received a technique of fascial stretching in the lumbar area while the control group participated in an off magnetotherapy machine. The hamstring flexibility in both lower limbs was measured by the Straight Leg Raising Test (SLR) and the Passive Popliteal Angle Test (PKE).

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 39 years old.
* Signed informed consent

Exclusion Criteria:

* Any alteration that prevents the normal communication between the patient and the therapist at the time of the study.
* Have an injury in the hamstring muscles.
* Have a chronic or acute lumbar pain in the moment of the realization.
* Neurological or orthopedic desease.
* Any important estructural alteration in the lower members that may be likely to alter the results under study.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Straight Leg Raising Test (SLR) | Pre-intervention and immediately after the intervention
  Test
Change from Passive Popliteal Angle Test (PKE) | Pre-intervention and immediately after the intervention
  Test

SECONDARY OUTCOMES:
IPAQ | Pre-intervention
  Cuestionnary

CONTACTS AND LOCATIONS:
Overall Officials: Juan Javier Bru Ruiz, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Spain